CLINICAL TRIAL: NCT00664118
Title: In Combination of Doula and Epidural Analgesia in the Latent Phrase of Labor in Primiparous Women
Brief Title: Doula Combined Latent Phrase Epidural Analgesia in Primiparous Women
Acronym: DCLEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMCHCH-0121-236; NMUC-08022
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Labor Pain
Keywords: Doula; Patient-controlled epidural analgesia; Neuraxial analgesia; Labor analgesia
MeSH Terms: conditions — Labor Pain | interventions — Analgesia; Doulas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Doula combined epidural analgesia in the latent phase of first stage of labor
  Interventions: Procedure: Doula combined analgesia
- 2 (Sham Comparator): Epidural analgesia in the latent phase of the first stage of labor without doula accompany
  Interventions: Procedure: Analgesia without doula

INTERVENTIONS:
Procedure: Doula combined analgesia — Doula combined epidural analgesia in the latent phase of first stage of labor in primiparas
  Arms: 1
Procedure: Analgesia without doula — Epidural analgesia in the latent phase of first stage of labor without doula accompany in primiparas
  Arms: 2

SUMMARY:
Accumulating evidence indicated that neuraxial analgesia in the latent phase of the first stage of labor would be an effective and safe health care procedure for nulliparas. Doulas, women with labor experience trained for parturients, is a new way to alleviate the psychological stress from the laboring pain. Previous data in our study showed that doula accompany is a good method in shortening the progress of labor used in the active phrase of the first stage of labor, and decreasing the rate of cesarean delivery. Investigators hypothesized that doula combined neuraxial (epidural) analgesia in the latent phrase would be a superior means for effective pain relief, decreased rate of cesarean section, and shortened duration of labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* > 18 years and < 45 years
* Spontaneous labor
* Analgesia request

Exclusion Criteria:

* Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records
* Participants younger than 18 years or older than 45 years
* Those who were not willing to or could not finish the whole study at any time
* Using or used in the past 14 days of the monoamine oxidase inhibitors;
* Alcohol addictive or narcotic dependent patients were excluded for their influence on the analgesic efficacy of the epidural analgesics
* Subjects with a nonvertex presentation or scheduled induction of labor
* Cervical dilation was 4.0 cm or greater before performing epidural puncture and catheterization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Rate of cesarean delivery | Analgesia initiation (0 h) to completion of vaginal delivery (4-7 h)

SECONDARY OUTCOMES:
Rate of instrumental delivery | Analgesia initiation (0 h) to successful vaginal delivery (4-7 h)
Indications of cesarean delivery | Analgesia initiation (0 h) to cesarean section (4-7 h)
Maternal Visual Analog Scale (VAS) rating of pain | 15 min prior to analgesia, 0-3 h of the latent phrase, 2-3 h of the active phrase, 1-2 h of the second stage of labor, 15 min posterior to delivery
Incidence of side effects | The whole period of the analgesia to successful vaginal delivery
Low back pain at 3 months after vaginal delivery | Three months after vaginal delivery
Maternal oral temperature | The whole period of the analgesia to successful vaginal delivery
Use of oxytocin after analgesia | During the whole period of the analgesia
Maximal oxytocin dose | 30 min after vaginal delivery
Duration of analgesia | Initiation of analgesia (0h) to the disappearance of sensory block (4-8h)
Breastfeeding success at 6 weeks after vaginal delivery | Six weeks after successful delivery
Maternal satisfaction with analgesia | 30 min after the vaginal delivery
Neonatal one-minute Apgar scale | One minute after baby was born
Neonatal five-minute Apgar scale | Five minutes after baby was born
Umbilical-cord gases analysis | Immediately after baby was born
Neonatal sepsis evaluation | 5 min after the baby was born
Neonatal antibiotic treatment | 5 min after the baby was born

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China